CLINICAL TRIAL: NCT07107646
Title: Investigating the Efficacy of Perceptual Learning in Blurred Gabor Discrimination Among Children With Low Myopia: An Exploratory Study
Brief Title: Exploring Perceptual Learning in Blurred Gabor Discrimination for Low-Myopic Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202504046RIND
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Visual Rehabilitation; Perceptual Learning
Keywords: Low Myopia; Perceptual Learning; Visual Acuity; Visual Evoked Potentials
MeSH Terms: conditions — Myopia | interventions — Tidal Volume

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Perceptual Learning Group (Experimental): Children aged 6-10 years with low myopia will receive a structured visual perceptual learning (VPL) intervention using computerized blurred Gabor discrimination tasks. Training will be conducted at least twice per week, with each session lasting approximately 15-30 minutes, for up to 3 months. Training parameters will be remotely monitored and adjusted based on individual progress. Participants will undergo baseline, post-training, and follow-up assessments of uncorrected visual acuity, refractive error, contrast sensitivity, visual crowding, Chinese reading visual acuity, eye movement performance, and sweep visual evoked potentials (sVEP).
  Interventions: Behavioral: vision training system, VTS
- Control Group (No Intervention): Children aged 6-10 years with low myopia who meet the same inclusion and exclusion criteria will not receive the VPL training during the study period. They will undergo the same schedule of baseline, post-study, and follow-up assessments as the experimental group, including evaluations of uncorrected visual acuity, refractive error, contrast sensitivity, visual crowding, Chinese reading visual acuity, eye movement performance, and sweep visual evoked potentials (sVEP).

INTERVENTIONS:
Behavioral: vision training system, VTS — Participants in this group will receive individualized visual perceptual learning using the Vision Training System (VTS). The training involves blurred Gabor stimuli presented via a computer-based application. Each participant will complete approximately 20 training sessions over 3 months, with each session lasting 15 to 30 minutes, conducted twice per week. The program is designed to enhance uncorrected visual acuity, contrast sensitivity, and other visual functions by engaging neural mechanisms related to perceptual learning. Training progression is adaptive based on individual performance. The VTS software was developed in collaboration with Bar Ilan University.
  Arms: Visual Perceptual Learning Group

SUMMARY:
This exploratory study investigates whether perceptual learning using blurred Gabor stimuli can improve uncorrected distance visual acuity in children aged 6-10 years with low myopia. Participants will be randomly assigned to a training group or control group. The training group will undergo individualized visual perceptual learning through a digital Vision Training System (VTS) for approximately 3 months. The study will also evaluate changes in refraction, contrast sensitivity, visual crowding, Chinese reading acuity with eye movements, and sweep visual evoked potentials (sVEPs).

DETAILED DESCRIPTION:
Perceptual learning (PL) is a non-invasive approach that enhances visual function through repeated visual tasks. Prior studies have demonstrated its potential in treating amblyopia and age-related visual decline. However, its application in children with low myopia remains underexplored.

This study has two main objectives:

To examine the effect of perceptual learning using blurred Gabor stimuli on uncorrected distance visual acuity in children with low myopia.

To investigate whether such training also improves refraction, contrast sensitivity, visual crowding, reading vision with eye movement patterns, and sweep visual evoked potentials (sVEPs).

Thirty children aged 6-10 years with spherical equivalent refractive errors between -0.50 and -1.25 diopters (including ≤ -0.75 diopters of astigmatism) will be enrolled. Participants will be randomized into a training group or control group. The training group will undergo approximately 20 sessions of individualized visual perceptual learning using the Vision Training System (VTS), developed in collaboration with Bar Ilan University.

Outcomes will be assessed before and after the intervention, and at follow-up points up to 12 months. Measures include visual acuity, refractive status, contrast sensitivity (CSV-1000E), crowding acuity (FrACT), Chinese reading visual acuity (with Tobii eye tracking), and sVEPs.

ELIGIBILITY:
Experimental and Control Group

Inclusion Criteria:

1. Children aged between 6 to 10 years.
2. Best corrected distance visual acuity of 6/6 or 0.00 logMAR.
3. Diagnosed with low myopia after a comprehensive ophthalmologic examination, with a spherical equivalent refractive error ranging from -0.50 to -1.25 diopters, including up to -0.75 diopters of astigmatism.
4. Not currently undergoing any of the four standard myopia control treatments for children:

   1. Atropine (mydriatic agent)
   2. Orthokeratology
   3. Peripheral defocus soft contact lenses
   4. Peripheral defocus spectacle lenses (frame glasses)
5. Willing and able to provide informed consent, and able to comply with study procedures and assessments.

Exclusion Criteria:

Participants will be excluded if they have any of the following ophthalmologic conditions:

1. Strabismus
2. Binocular vision problems
3. Ocular diseases
4. History of ocular surgery (excluding refractive surgery)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) From Baseline | From enrollment to 12 months after completion of the 3-month training program
  Best Corrected Visual Acuity (BCVA) will be measured using the ETDRS or Snellen chart at a distance of 3 meters under standardized lighting conditions. The change in BCVA from baseline to post-training will be assessed.

SECONDARY OUTCOMES:
Change in Spherical Equivalent Refraction (Diopters) From Baseline | From enrollment to 12 months after completion of the 3-month training program
  Spherical equivalent refraction will be measured using both automated and subjective refraction methods. Changes in spherical equivalent diopters will be assessed and compared between groups.
Change in Contrast Sensitivity Across Spatial Frequencies From Baseline | From enrollment to 12 months after completion of the 3-month training program
  Contrast sensitivity will be measured using the CSV-1000E test at a distance of 2.5 meters, assessing spatial frequencies at 3, 6, 12, and 18 cycles per degree (cpd). Changes from baseline will be evaluated.
Change in Visual Crowding Acuity From Baseline | From enrollment to 12 months after completion of the 3-month training program
  Visual crowding acuity will be assessed using the Freiburg Vision Test (FrACT) before and after the training program. Changes from baseline will be evaluated.
Change in Reading Visual Acuity and Eye Movement Parameters From Baseline | From enrollment to 12 months after completion of the 3-month training program
  Reading visual acuity and eye movements will be assessed using a custom Chinese reading test for children. Eye movements will be recorded using a Tobii eye tracker. Measured metrics include critical print size, maximum reading speed, and maximum reading acuity. Changes from baseline will be evaluated.
Change in Visual Acuity Measured by Sweep Visual Evoked Potentials (sVEP) From Baseline | From enrollment to 12 months after completion of the 3-month training program
  Objective visual acuity will be measured using the sweep visual evoked potentials (sVEP) technique. Neural responses will be compared between pre- and post-training assessments to evaluate changes in visual acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Occupational Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No